CLINICAL TRIAL: NCT05179538
Title: Laying the Groundwork for Personalized Medicine in Aphasia Therapy: Genetic and Cognitive Predictors of Restorative Treatment Response
Brief Title: Genetic and Cognitive Predictors of Aphasia Treatment Response
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60066189
Record Dates: First submitted 2021-08-25; First posted 2022-01-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: There will be four subgroups based on the expression of BDNF and ApoE.
Masking Description: Speech-language pathologists who will be providing assessments and therapy will be blinded to participant genotypes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Treatment (Experimental): Cued picture naming therapy will be delivered to all participants. There will be four cohorts of participants based on BDNF and ApoE genotypes.
  Interventions: Behavioral: Cued picture-naming therapy

INTERVENTIONS:
Behavioral: Cued picture-naming therapy — The proposed study will administer Cued Picture-Naming Treatment (CPNT) four days per week for four weeks (i.e. 16 sessions). During therapy, participants will attempt to name eight consecutive presentations of the same black and white picture, for each of the 20 pictures, with cueing from the administrator. Trials will include (1) independent naming, (2) orthographic cueing (i.e. the written word beneath the picture.), (3) repeating, (4) naming after a short delay (i.e. approximately three seconds), (5)semantic cueing (i.e. three cues providing semantic information about the target will be spoken to the participant by the clinician), (6) phonological cueing (i.e. the first sound and letter will be spoken by the clinician), (7) repeating, and (8) naming after a short delay. The administrator will provide the correct response for each incorrect participant response and will ask the participant to repeat it.

SUMMARY:
Aphasia, or language impairment after a stroke, affects approximately 2 million people in the United States, with an estimated 180,000 new cases each year. The medical community cannot predict how well someone with aphasia will respond to treatment, as some people with aphasia are poor responders to intervention even when participating in empirically supported treatments. There is a strong likelihood that genetics play a role in language recovery after stroke, but very little research has been dedicated to investigating this link. This study will investigate whether two genes and cognitive abilities, such as memory, predict responsiveness to aphasia therapy for word-retrieval difficulties.

DETAILED DESCRIPTION:
Incomplete understanding of patient-specific factors that determine whether someone will respond well to language therapy after stroke limits the development of methods to target or account for sources of variability. There is a strong likelihood that genetics play a role in language recovery after stroke, but very little research has been dedicated to investigating this link. The long-term goal of this line of work is to maximize response to aphasia therapy by incorporating patient-specific factors into decisions related to treatment planning. The overall objective of this application is to identify patterns of patient-specific factors including two candidate genes and cognitive skills that show a relationship with treatment outcomes. The central hypothesis is that there will be a relationship between ApoE and BDNF genotypes, and working memory on stimulus generalization. The rationale for the proposed project is that the identification of factors that impact treatment responsiveness will allow for better estimation of prognosis, improved triage of individuals into appropriate therapy regimens and direct targeting of cognitive factors to maximize behavioral gains. The two specific aims of the project are to determine the degree to which (1) ApoE and BDNF genotypes influence how individuals with aphasia respond to therapy, and (2) working memory abilities are related to stimulus acquisition and stimulus generalization after anomia therapy. Individuals with chronic post-stroke aphasia will undergo cognitive and language assessment, and provide a saliva sample for genetic analysis prior to participating in a cued picture-naming therapy for anomia. The expected outcomes are to integrate cognitive scores and genotypes for BDNF and ApoE into formulating probabilities of individual patient responsiveness to restorative therapy. Improvement in word retrieval abilities will be evaluated using the percentage of pictures named correctly. This contribution is expected to be significant because it will allow for more informed clinical decision making and better allocation of resources to appropriate treatments, thereby making advances in the field toward more personalized medicine, as opposed to a one-size-fits-all clinical approach.

The investigators will determine genotypes for BDNF and ApoE, which will yield four separate groups. At least 20 participants will be enrolled for each genotype group.

ELIGIBILITY:
Inclusion Criteria:

* At least six months post-onset of a single left-hemisphere stroke
* Chronic aphasia
* Anomia (word-retrieval deficits)
* Native English Speaker.

Exclusion Criteria:

* Severe motor speech disorders
* Severe auditory comprehension deficits
* Severe depression.
* Diffuse injury or disease of the brain
* Uncorrected vision or hearing difficulties
* Contraindications for MRI (e.g. cardiac pacemaker, ferrous metal implants, claustrophobia, pregnancy).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent of pictures named correctly | from baseline to 1 month
  Picture-naming score changes from baseline to post-treatment.
Percentage of pictures named correctly | 4 months
  Picture-naming score changes from post-treatment to follow up.

SECONDARY OUTCOMES:
percentage of definitions named correctly | after 1 month
  Changes in naming pictures trained from definition from baseline to post-treatment
Percentage of untrained pictures named correctly | after 1 month
  Changes in naming of untrained items from baseline to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stacy M Harnish, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No